CLINICAL TRIAL: NCT03442010
Title: Incidence and Risk Factor of Adverse Drug Events Detected at Emergency Department Visit
Brief Title: Adverse Drug Events at Emergency Department
Acronym: ADEsED
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0095
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Adverse Drug Event
Keywords: Emergency department; Clinical Pharmacist; Adverse drug event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with adverse drug event: People with adverse drug event
  Interventions: Other: Detection of adverse drug events
- People without adverse drug event: People without adverse drug event

INTERVENTIONS:
Other: Detection of adverse drug events — Detection of adverse drug events
  Groups: People with adverse drug event

SUMMARY:
Emergency departments (EDs) are a crucial element of the health care systems at interface between hospital and communities. The goals of the ED are to make an initial diagnosis and deliver urgent and critical care 24 hour per day and 365 days a year. Also, many Adverse Drug Events (ADEs) are not identified by emergency physicians. ADEs are injuries resulting from a drug related medical intervention. Their detection, documentation and reporting are essential for adequate medical care and knowledge of risk/benefit profiles of medication throughout their lifecycle. However, a number of studies indicate that in clinical practice the under-reporting of ADEs is a pervasive and widespread problem. The main reasons for under-reporting were difficulty in determining the cause of the ADE, lack of time, poor integration of ADE-reporting systems and uncertainty about reporting procedures. Successful treatment of ADEs depends on the ability of physicians to attribute ADEs to a medication. Some studies have reported that pharmacists but also student pharmacists were one of the best health care providers to establish medication history. Consequently, the aims of our study were to assess prevalence and characteristics of ADEs identified in an emergency department and to identify factors associated with ADEs in ED patients.

This prospective observational study is conducted at the ED of a tertiary care hospital (University hospital of Montpellier). This department supports 80 000 patients every years. Patient were not included if they were less than 18 years old, present acute psychological disturbance or they did not agree to participate at this study.

For each patient included, a pharmaceutical team conducted: medication reconciliation process to establish medication history and a structured interviews to determine self-reported adherence and self-medication. ADEs were attributed to a medication by the treating senior emergency physician: directly during patient consultation or after being alerted by the pharmaceutical team.

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the department during the study period

Exclusion criteria:

- Patient presenting acute psychological disturbance or they did not agree to participate at this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient admitted in emergency department of Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 13453 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug events | 1 day
  Number of adverse drug events identified in a emergency deparmtent

SECONDARY OUTCOMES:
number of variable associated with adverse drug events | 1 day
  number of variable associated with adverse drug events in ermergency department patients

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Lohan L, Marin G, Faucanie M, Laureau M, Macioce V, Perier D, Pinzani V, Giraud I, Castet-Nicolas A, Jalabert A, Villiet M, Sebbane M, Breuker C. Impact of medication characteristics and adverse drug events on hospital admission after an emergency department visit: Prospective cohort study. Int J Clin Pract. 2021 Jul;75(7):e14224. doi: 10.1111/ijcp.14224. Epub 2021 Apr 23. PMID 33866662
- [Derived] Laureau M, Vuillot O, Gourhant V, Perier D, Pinzani V, Lohan L, Faucanie M, Macioce V, Marin G, Giraud I, Jalabert A, Villiet M, Castet-Nicolas A, Sebbane M, Breuker C. Adverse Drug Events Detected by Clinical Pharmacists in an Emergency Department: A Prospective Monocentric Observational Study. J Patient Saf. 2021 Dec 1;17(8):e1040-e1049. doi: 10.1097/PTS.0000000000000679. PMID 32175969